CLINICAL TRIAL: NCT03091270
Title: The Application of ZOOMit-fMRI to Identify Motor Functional Cortex
Brief Title: ZOOMit-fMRI Identifies Motor Functional Cortex
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: NSFC-81601452
Record Dates: First submitted 2017-03-16; First posted 2017-03-27 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Gliomas
Keywords: gliomas; motor functional cortex; ZOOMit-fMRI; BOLD-fMRI
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (2):
- BOLD-fMRI: Identifying the motor functional cortex in glioma patients with BOLD-fMRI.
- ZOOMit-fMRI: Identifying the motor functional cortex in glioma patients with ZOOMit-fMRI.

SUMMARY:
This study was designed to collect a series of patients with gliomas which were involved in motor cortex to analyze difference accuracy of motor cortex localization between BOLD-fMRI and ZOOMit-fMRI.

DETAILED DESCRIPTION:
Gliomas will lead motor dysfunction when they are involved in motor cortex. However, tumor resection also have risk to lead postoperatively motor function deficits if destroy patients' motor cortex when tumor removed. Hence, it is important for neurosurgeon to realize the situation of patients' motor cortex locations in order to determine personal operative protocol.

The blood oxygen level dependent fMRI (BOLD-fMRI) is a prevalent preoperative method to localization motor cortex. It shows motor relevant cortex by the change of blood oxygen level when patients cooperate to finish motor tasks. The advantage of BOLD-fMRI includes higher time and spatial resolution, higher sensitivity, non-invasive. However, its accuracy of localization has not been satisfactory because neurovascular uncoupling. The ZOOMit-fMRI is a novel technic which is evolved from conventional BOLD-fMRI to localize motor functional cortex.The advantage of ZOOMit-fMRI is smaller field of view (FOV) and higher spatial resolution comparing with BOLD-fMRI. That helps to reduce other region of brain interference and elevate accuracy of localizations.

In this study, the investigators plan to enroll 60 patients, whose gliomas are involved in motor cortex, to acquire their BOLD-fMRI and ZOOMit-fMRI data in order to analyze their difference in the accuracy of motor cortex localization.

ELIGIBILITY:
The inclusion criteria were as follows: 1) age ≥ 18 years; 2) no history of surgical treatment or radiotherapy; 3) no contraindication to MRI scanning; 4) agreeable to receive the fMRI scanning and awake craniotomy with DCS.

The exclusion criteria were as follows: 1) basing on the anatomic MRI, the distance from the tumor to the hand-knob area lower than 20 mm; 2) disable to finish the task of clenching fist during fMRI scanning.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with gliomas which are closed to motor area (including primary motor area, premotor area and supplementary area), treated by awake craniotomy and intraoperative brain mapping
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The accurate rate for hand motor cortex localization with BOLD-fMRI and ZOOMit-fMRI. | From scanning with BOLD-fMRI and ZOOMit-fMRI to getting the overlap indexes,assessed up to 2 weeks in each patient.
  To illustrate the accurate rate of hand motor cortex localization, the overlap indexes in BOLD-fMRI or ZOOMit-fMRI will be calculated. The results in BOLD-fMRI and ZOOMit-fMRI will be defined with 300 maximum value voxels via Statistical Parametric Mapping 8 (SPM8) software. According to the photographs and records of direct cortical stimulation (DCS) during awaken craniotomy, the DCS results will be confirmed as a global region with 5 mm diameter. Subsequently, we will overlap the BOLD-fMRI/ZOOMit-fMRI and DCS results then calculate the number of voxels overlapping. In this way, the overlap indexes can be calculated as a ratio between the number of voxels overlapping and the number of total voxels in BOLD-fMRI and ZOOMit-fMRI. We defined if the overlap index is larger than 0, the localization result is accurate. In contrast, if the overlap index is equal to zero, the localization result is inaccurate. Finally, the accurate rate of hand motor cortex localization can be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Neurosurgical Institute and Beijing Tiantan Hospital, Beijing, Beijing Municipality, China